CLINICAL TRIAL: NCT01877447
Title: Comparison of Two Transcranial Direct Current Stimulation (tDCS) Protocols for the Treatment of Major Depressive Disorder: a Randomized, Double-blinded, Controlled Clinical Trial.
Brief Title: Comparison of Two tDCS Protocols for the Treatment of Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Andre Brunoni, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: aF3_cF4_F32
Record Dates: First submitted 2013-05-24; First posted 2013-06-13 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: MAjor Depressive Disorder
Keywords: tDCS; Brain stimulation; depressive disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder | interventions — Transcranial Direct Current Stimulation; Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cathodal F4 (Experimental): Transcranial Direct Current Stimulation
  Cathodal tDCS over F4 (right dorsolateral prefrontal cortex) Anodal tDCS over the left deltoid (extra-cephalic) n=15
  Interventions: Device: Transcranial Direct Current Stimulation
- Anodal F3 (Experimental): Transcranial Direct Current Stimulation'
  Anodal tDCS over F3 (right dorsolateral prefrontal cortex) Cathodal tDCS over the right deltoid (extra-cephalic) n=15
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Current Stimulation with cathodal stimulation over right dorsolateral prefrontal cortex. Anodal stimulation over left deltoid region
  Other Names: tDCS; Brain polarization; Brain stimulation

SUMMARY:
Transcranial direct cranial stimulation (tDCS) is a novel technique based on the application of a weak electrical current over the scalp through two electrodes - the anode, which facilitates neuronal depolarization, and the cathode, which leads to neuronal hyper-polarization. Recently, several open-label and sham-controlled clinical trials applied daily tDCS sessions for the treatment of major depressive disorder (MDD). Theoretically, tDCS displays depression improvement through anodal stimulation over the left dorsolateral prefrontal, inducing excitability-enhancing effects over this area, which is hypoactive during the acute depressive episode. The present study is aimed at comparing two different tDCS protocols: (1) active anodic stimulation over left dorsolateral prefrontal cortex with cathode placed over an extra cephalic area; (2) active cathode placed over the right dorsolateral prefrontal cortex with anode placed over an extra cephalic area.

DETAILED DESCRIPTION:
The present research protocol will evaluate clinical effects of two different tDCS protocols: (1) active anodic stimulation over left dorsolateral prefrontal cortex with cathode placed over an extra cephalic area; (2) active cathode placed over the right dorsolateral prefrontal cortex with anode placed over an extra cephalic area. Patients will be clinically evaluated with the Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria for depression. Symptoms intensity will be rated according to The Hamilton Depression Scale (HAMD -17 items) - main outcome. Patients with scores higher than 16 will be included. Patients with active neurological or severe disorders (such as cancer or auto-imune disorders) will be excluded. The present study is a double-blinded, controlled, randomized trial with 30 patients with depression. The intervention protocol consist in 15 consecutive daily tDCS sessions (skipping the weekend). After meeting eligibility criteria, patients will be randomized (computer generated list) to one of the two intervention groups. We will use a direct current of 2.0 milliamperes (mA) for 30 min. The 35 cm2-rubber electrodes will be wrapped in cotton material, which should be moistened with saline as to reduce impedance. Patients will be clinically assessed at baseline and at end of 6 weeks. Main outcome will be based on HAMD-17 items at a final endpoint of 6-weeks, with secondary outcomes assessing Beck Depression Inventory (21 items) at 6 weeks. Other evaluation scales include Beck Anxiety Inventory, Hamilton Anxiety Scale and Safety and cognitive assessment will be performed with The Montreal Cognitive Assessment, adverse effects scales and clinical evaluation with a trained physician.

ELIGIBILITY:
Inclusion Criteria:

* patients with age between 18-89 years, depression diagnosis according to Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-iV); HAMD scores higher than 16; accordance to inform consent

Exclusion Criteria:

* active neurologic or severe disorder (such as cancer or auto-imune)
* pregnancy;
* need for hospitalization

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression, 17 items (HAMD17) | Weeks 0, 3 and 6
  reduction of depressive symptoms as assessed by HAMD17

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Weeks 0, 3 and 6
  reduction of depressive symptoms as assessed by MADRS
Beck Depression Inventory (BDI) | Weeks 0, 3 and 6
  reduction of depressive symptoms as assessed by BDI
Beck Anxiety Inventory (BAI) | Weeks 0, 3 and 6
  reduction of anxiety symptoms as assessed by BAI
Hamilton Anxiety Inventory (HAI) | Weeks 0, 3 and 6
  reduction of anxiety symptoms as assessed by HAI
The Montreal Cognitive Assessment (Moca) | Weeks 0 and 6
  evaluate cognitive stability as assessed by Moca

CONTACTS AND LOCATIONS:
Overall Officials: Andre R Brunoni, PhD, Principal Investigator — Center of Clinical Research - Hospital Universitário USP; Sao Paulo; Brazil
Locations (1):
- Hospital Universitário - USP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Brunoni AR, Kemp AH, Shiozawa P, Cordeiro Q, Valiengo LC, Goulart AC, Coprerski B, Lotufo PA, Brunoni D, Perez AB, Fregni F, Bensenor IM. Impact of 5-HTTLPR and BDNF polymorphisms on response to sertraline versus transcranial direct current stimulation: implications for the serotonergic system. Eur Neuropsychopharmacol. 2013 Nov;23(11):1530-40. doi: 10.1016/j.euroneuro.2013.03.009. Epub 2013 Apr 21. PMID 23615118
- [Background] Brunoni AR, Benute GR, Fraguas R, Santos NO, Francisco RP, de Lucia MC, Zugaib M. The self-rated Inventory of Depressive Symptomatology for screening prenatal depression. Int J Gynaecol Obstet. 2013 Jun;121(3):243-6. doi: 10.1016/j.ijgo.2013.01.011. Epub 2013 Mar 15. PMID 23499135
- [Background] Kalu UG, Sexton CE, Loo CK, Ebmeier KP. Transcranial direct current stimulation in the treatment of major depression: a meta-analysis. Psychol Med. 2012 Sep;42(9):1791-800. doi: 10.1017/S0033291711003059. Epub 2012 Jan 12. PMID 22236735
- [Background] Brunoni AR, Valiengo L, Baccaro A, Zanao TA, de Oliveira JF, Goulart A, Boggio PS, Lotufo PA, Bensenor IM, Fregni F. The sertraline vs. electrical current therapy for treating depression clinical study: results from a factorial, randomized, controlled trial. JAMA Psychiatry. 2013 Apr;70(4):383-91. doi: 10.1001/2013.jamapsychiatry.32. PMID 23389323
- [Background] Brunoni AR, Ferrucci R, Fregni F, Boggio PS, Priori A. Transcranial direct current stimulation for the treatment of major depressive disorder: a summary of preclinical, clinical and translational findings. Prog Neuropsychopharmacol Biol Psychiatry. 2012 Oct 1;39(1):9-16. doi: 10.1016/j.pnpbp.2012.05.016. Epub 2012 May 28. PMID 22651961
- [Background] Brunoni AR, Ferrucci R, Bortolomasi M, Vergari M, Tadini L, Boggio PS, Giacopuzzi M, Barbieri S, Priori A. Transcranial direct current stimulation (tDCS) in unipolar vs. bipolar depressive disorder. Prog Neuropsychopharmacol Biol Psychiatry. 2011 Jan 15;35(1):96-101. doi: 10.1016/j.pnpbp.2010.09.010. Epub 2010 Sep 18. PMID 20854868